CLINICAL TRIAL: NCT07085780
Title: A Prospective, Open-Label, Single-Centre Interventional Study to Evaluate the Efficacy and Safety of Dharasana Lep in Patients With Mild to Moderate Musculoskeletal Pain and Rheumatoid Arthritis.
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Dharasana Lep in Patients With Mild to Moderate Muscular, Joint, or Rheumatic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Shah Maganlal Chunilal Gandhi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB250029-SM
Record Dates: First submitted 2025-07-09; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Pain; Rheumatic Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dharasena Pain Relief Lep (Experimental): 1. Apply a thin, even layer of the Lep directly onto the clean and dry affected area.
  2. Cover the application with a layer of clean cotton.
  3. Allow the Lep to remain on the area for at least 2 days,
  4. Avoiding exposure to direct heat or open flame during this period.
  5. In this study, on Day 04, gently remove the Lep using warm water and soft cotton cloth and thoroughly cleanse the area with mild soap and water.
  Interventions: Other: LEP

INTERVENTIONS:
Other: LEP — 1. Apply a thin, even layer of the Lep directly onto the clean and dry affected area.
  2. Cover the application with a layer of clean cotton.
  3. Allow the Lep to remain on the area for at least 2 days,
  4. Avoiding exposure to direct heat or open flame during this period.
  5. In this study, on Day 04, gently remove the Lep using warm water and soft cotton cloth and thoroughly cleanse the area with mild soap and water.

SUMMARY:
A Prospective, Open-Label, Single-Centre Interventional Study to Evaluate the Efficacy and Safety of Dharasana Lep in Patients with Mild to Moderate Musculoskeletal Pain and Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is an open-label, single-centre, prospective, interventional, clinical study to evaluate the efficacy and safety of pain relief lep in patients with mild to moderate musculoskeletal pain and rheumatoid arthritis. A total of 35 participants will be enrolled in the study, including males and non-pregnant, non-lactating females aged between 25 and 65 years (inclusive). Participants experiencing musculoskeletal pain of mild to moderate intensity, such as knee pain, swelling, back pain, muscle sprains, or strains will be enrolled in the study. Among the total, 5 participants will have a diagnosis of Rheumatoid Arthritis with associated walking difficulty. The study aims to complete with 30 evaluable participants, accounting for potential dropouts or withdrawals during the study period.

The potential subjects will be screened as per the inclusion and exclusion criteria only after obtaining the written informed consent from the study participants. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by recruiting department prior the enrolment visit. During the screening process (prior to enrolment), participants will be instructed to refrain from using any other topical analgesics or pain relief medications before and throughout the study period.

There will be a total of 2 visits during the study - Visit 01 (01 Day) and Visit 02 (04 Day). The duration of the study will be 04 Days (2 Days) from the enrolment. Subjects will be instructed to visit the facility as per below visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25-65 years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Subject is in good general health as determined by the Investigator on the basis of medical history.
4. Subject must be having presence of body ache, joint or muscle pain, sprain/strain, or back pain for more than 1 week and less than 6 months.
5. Patients must have a confirmed diagnosis of mild to moderate musculoskeletal pain and rheumatic conditions with a pain score between 4 - 7, grade will be evaluated using Visual Analog Scale (VAS).
6. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
7. If the subject is of childbearing potential they must have a self-reported negative urine pregnancy, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
8. Subjects are willing to give written informed consent and are willing to follow the study procedure.
9. Subjects who commit not to use any other medicated/ prescription topical analgesics or medication, other than the test treatment for the entire duration of the study.
10. Subject is willing and able to comply with study procedures, including all scheduled visits, treatment applications, and assessments.
11. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
12. Subject must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Subject has severe arthritis requiring prescription medication including immunomodulators, COX Inhibitors, etc.
2. Subjects having any skin disorder or presence of open wounds, cut, bruising, rashes etc.
3. Subjects with raw wounds, sutures, fractures and hematoma.
4. Subjects suffering from auto-immune disorder, spastic disorder, genetic disorder and any other sever traumatic conditions.
5. Subjects with chronic pain like arthritis, gout, and ankylosing spondylitis.
6. Subject have history of any hypersensitivity to the ingredients in the Lep.
7. Subject who had taken any systemic product for any illnesses for at least 3 months.
8. History of alcohol or drug addiction.
9. Pregnant or breast feeding or planning to become pregnant during the study period.
10. History of chronic illness which may influence the cutaneous state.
11. Subject have participated any clinical research study within the last 30 days.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in Pain Intensity evaluated through Visual Analogue Scale (VAS) | From baseline prior to application of test treatment on Day 01, telephonic follow up on Day 02 and post removal of test treatment on Day 04 (+2 Days).
  The Visual Analogue Scale is a 10 point scale. In which 0 means no pain and 10 means severe pain.

SECONDARY OUTCOMES:
Improvement in Joint stiffness and movement evaluated through Numeric Pain Rating Scale (NPRS) | From baseline prior to application of test treatment on Day 01, and post removal of test treatment on Day 04 (+2 Days).
  The Numeric Pain Rating Scale is a 10 point scale. In which 0 means no pain and 10 means severe pain.
Improvement in flexibility / extent of movement of joint evaluated through Range of Motion (ROM) assessment | From baseline prior to application of test treatment on Day 01, and post removal of test treatment on Day 04 (+2 Days).
Improvement in Vedana assessment and management evaluated through Ayurvedic Pain Assessment and Management scale (APMS) | From baseline prior to application of test treatment on Day 01, and post removal of test treatment on Day 04 (+2 Days).
Improvement in aggravated doshas (Vata, Pitta, Kapha) evaluated through ayurvedic clinical examination | From baseline prior to application of test treatment on Day 01, and post removal of test treatment on Day 04 (+2 Days).
  Improvement in aggravated Doshas (Vata, Pitta, Kapha) will be assessed using a standardized Ayurvedic clinical examination scale, based on classical signs and symptoms. Each Dosha will be graded on a 4-point scale (0-3) indicating severity from absent to severe.
Improvement in product perception questionnaire using quality of life questionnaire through 5-point Likert scale to evaluate the changes in pain intensity, joint movement, stiffness, musculoskeletal pain and inflammation post treatment and PGIC scale | From baseline prior to application of test treatment on Day 01, and post removal of test treatment on Day 04 (+2 Days).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan Patel, Principal Investigator — NovoBliss Research Private Limited

IPD SHARING:
Plan to Share IPD: No